CLINICAL TRIAL: NCT04705740
Title: Influence of the Endoscopist Case Volumen on Endoscopic Retrograde CholangioPanceratography Outcomes
Brief Title: Influence of the Endoscopists and Endoscopic Retrograde CholangioPanceratography
Status: Completed | Type: Observational
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: NER20
Record Dates: First submitted 2020-12-11; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Biliary Disease; Pancreatic Diseases
Keywords: ERCP; endoscopy; gastrointestinal; choledocholithiasis; Endoscopic Retrograde CholangioPanceratography
MeSH Terms: conditions — Gallbladder Diseases; Pancreatic Diseases; Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- September 2013 to August 2015: 5 endoscopists
  Interventions: Other: ERCP
- September 2015 to December 2017: 4 endoscopists
  Interventions: Other: ERCP
- January 2018 to June 2020: 3 endoscopists
  Interventions: Other: ERCP

INTERVENTIONS:
Other: ERCP — ERCPs performed annually by an endoscopist

SUMMARY:
Retrospective analysis on a prospective database that analyzes the influence of the number of endoscopists on the Endoscopic Retrograde CholangioPanceratography result.

DETAILED DESCRIPTION:
The number of Endoscopic Retrograde CholangioPanceratographys (ERCP) performed annually by an endoscopist has been shown to influence the outcomes of the procedure, especially on the papillary cannulation rate and the adverse effects rate. The number of ERCPs performed annually by each endoscopist is directly related to the number of endoscopists who perform this procedure, since the total number of ERCPs performed annually at each center is usually constant.

The hypothesis of this study is that the number of endoscopists who perform ERCP in a hospital influences the results of the procedure, so that the fewer the number of endoscopists the better the results.

To evaluate this hypothesis, the investigators have designed a retrospective study analyzing data from a prospectively filled database, which includes all ERCPs performed in our center from September 2013 to June 2020. For organizative reasons unrelated to the endoscopy unit, in the center it has beed progressively reduced the number of endoscopists who perform ERCP, starting from 5 endoscopists at the beginning of the study to 3 endoscopists at the end of the study inclusion period. In fact, three different periods of similar duration can be distinguished: September 2013 to August 2015 (5 endoscopists), September 2015 to December 2017 (4 endoscopists) and January 2018 to June 2020 (3 endoscopists).

The outcomes obtained with ERCP in these three periods will be analyzed and compared, assessing the cannulation rate and the adverse effects rate as the main comparison parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ERCP with written informed consent given
* Staff allocated in the endoscopy unit

Exclusion Criteria:

* Rejection to participate in the study
* ERCP procedures performed by fellows in training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, undergoing ERCP by the staff allocated in the endoscopy unit.
Sampling Method: Non-Probability Sample
Enrollment: 2561 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Papillary cannulation | During the procedure
  Rate of papillary cannulation.Success in achieving transpapillary access to the bile duct.It has to be confirmed fluoroscopically
Adverse effects | Up to 1 month after intervention
  Rate of adverse effect assessed by the ASGE classification

SECONDARY OUTCOMES:
Individual adverse effects | Up to 1 month after intervention
  Rate of individual adverse effect during the intervention
Complexity level of ERCP | During the ERCP procedure
  Complexity level of ERCP according to ASGE classification of complexity of the endoscopic procedures
Therapeutics performed with ERCP | During the ERCP procedure
  Techniques used during ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Vila, PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No